CLINICAL TRIAL: NCT06910098
Title: Assessment of Impact of Rosuvastatin Doses on Low Density Lipoprotein Levels, Creatinine Phosphokinase Levels and Aspartate Aminotransferase Levels: A Randomized Controlled Trail
Brief Title: Impact of Rosuvastatin Doses on LDL Levels, CPK Levels and Aspartate Aminotransferase Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Park Medical College (Other)
Responsible Party: Principal Investigator, Mirza Zeeshan Sikandar, Dr, Central Park Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHRF/RCT/238
Record Dates: First submitted 2025-03-22; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: LDL - Low Density Lipoprotein Receptor Disorder; Rosuvastatin
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): receiving drug dose of 5mg
  Interventions: Drug: Rosuvastatin
- Group 2 (Active Comparator): receiving grug dose of 10 mg
  Interventions: Drug: Rosuvastatin
- Group 3 (Active Comparator): receiving dose of 20 mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — a dose of 5mg were given and were compared for the cpk, ast and ldl levels
  Arms: Group 1
Drug: Rosuvastatin — a dose of 10 mg were given and were compared for the cpk, ast and ldl levels
  Arms: Group 2
Drug: Rosuvastatin — a dose of 20 mg were given and were compared for the cpk, ast and ldl levels
  Arms: Group 3

SUMMARY:
Particpants were divided into groups based on doses of rosuvastatin and were assessed and for CPK, LDL and AST levels

ELIGIBILITY:
Inclusion Criteria:

patients who were already on statins

Exclusion Criteria:

hereditary diseases including familial hypercholesterolemia and kidney diseases

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
impact of rosuvstatin over LDL, CPK and AST levels | 12 weeks
  Pre- and post intervention levels of fasting serum low-density lipoprotein (LDL) in mg/dL were recorded and were compared in all study groups for assessment of the impact of various doses of rosuvastatin.
impact of rosuvstatin over LDL, CPK and AST levels | 12 weeks
  Pre- and post-intervention levels of creatine phosphokinase (CPK) in mcg/L were recorded and were compared in all study groups for assessment of the impact of various doses of rosuvastatin in terms of rhabdomyolysis.
impact of rosuvstatin over LDL, CPK and AST levels | 12 weeks
  Pre- and post-intervention levels of Aspartate Aminotransferase (AST) in U/L were recorded and were compared in all study groups for assessment of the impact of various doses of rosuvastatin in terms of liver damage.

CONTACTS AND LOCATIONS:
Overall Officials: Sikandar, Principal Investigator — Central Park Medical College; Sikandar, Principal Investigator — Central Park Medical College & Teaching Hospital
Locations (1):
- Central Park Teaching Hospital, Lahore, Pakistan